CLINICAL TRIAL: NCT03306225
Title: Characterization of Endocarditis to Streptococci and Impact of the CMI on the Future of the Patients
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOSTREPTO
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Endocarditis, Bacterial
MeSH Terms: conditions — Endocarditis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The infectious endocarditis is a grave infection the incidence of which is at present esteemed at 30-100 episodes by million inhabitants a year.

This infection is marked with a heavy morbi-mortality.Preliminary studies seem to show an abnormally high death rate at the patients presenting an infectious endocarditis to streptococci with an inhibitive minimal concentration raised to the amoxicilline. The aim of the study is to describe the epidemiology and the clinical presentations of the patients presenting an endocarditis to streptococci

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* endocartitis with steptococci with Duke's criteria

Exclusion Criteria:

* age < 18 years
* suspiscious endocarditis without Duke's criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient diagnostised for endocarditis between 2010 and 2015
Sampling Method: Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of factors associated to the mortality in the patients presenting an endocarditis to streptococci. | an average of one year

CONTACTS AND LOCATIONS:
Overall Officials: PILMIS P Benoit, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France